CLINICAL TRIAL: NCT04731740
Title: Pembrolizumab in Combination With Standard 1st Line Therapy (Lenvatinib / Chemotherapy) for Locally Advanced or Metastatic Poorly Differentiated or Anaplastic Thyroid Cancer
Brief Title: Pembrolizumab and Lenvatinib/Chemotherapy for Poorly Differentiated/Anaplastic Thyroid Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Saint Petersburg State University, Russia (Other)
Responsible Party: Principal Investigator, Efremov Sergey, Principal Investigator, Saint Petersburg State University, Russia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 73
Record Dates: First submitted 2021-01-26; First posted 2021-02-01 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Metastatic Thyroid Gland Carcinoma; Poorly Differentiated Thyroid Gland Carcinoma; Thyroid Gland Anaplastic Carcinoma by AJCC V8 Stage
MeSH Terms: conditions — Thyroid Neoplasms | interventions — lenvatinib; pembrolizumab; Drug Therapy

STUDY DESIGN:
Intervention Model Description: Two parallel arms based on the inclusion/exclusion criteria: Pembrolizumab+Lenvatinib or Pembrolizumab+Chemotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pembrolizumab + Lenvatinib (Experimental): Experimental treatment:
  Lenvatinib p.o. once a day, pembrolizumab 200 mg i.v. every 21 days started 21 days after start of Lenvatinib
  Duration of treatment per patient:
  until the end of month 36 after registration of the last patient or disease progression or toxicity (whichever occurs first)
  Interventions: Drug: Lenvatinib; Biological: Pembrolizumab
- Pembrolizumab + Chemotherapy (Experimental): Experimental treatment:
  Investigators' choice of the Сhemotherapy, pembrolizumab 200 mg i.v. every 21 days started 21 days after the start of chemotherapy
  Duration of treatment per patient:
  until the end of month 36 after registration of the last patient or disease progression or toxicity (whichever occurs first)
  Interventions: Biological: Pembrolizumab; Drug: Chemotherapy

INTERVENTIONS:
Drug: Lenvatinib — PO
  Other Names: E7080; ER-203492-00
  Arms: Pembrolizumab + Lenvatinib
Biological: Pembrolizumab — IV
  Other Names: Keytruda; MK-3475; Lambrolizumab; SCH 900475
Drug: Chemotherapy — Investigators' choice
  Arms: Pembrolizumab + Chemotherapy

SUMMARY:
The aim of the study is to evaluate the efficacy of the combination of lenvatinib with pembrolizumab, and to establish a safe and effective systemic treatment regimen for patients with metastatic anaplastic thyroid cancer (ATC) / poorly differentiated thyroid cancer (PDTC).

Lenvatinib is an anti-angiogenic and antiproliferative drug used in differentiated thyroid cancer. It blocks proliferative genes such as RET and PDGFR and further inhibits major proliferation pathways such as VEGF receptor signaling and FGFR1-4.

Pembrolizumab is an immune checkpoint inhibitor that targets PD-1 located on lymphocytes. The response to pembrolizumab treatment is associated, among other things, with increased expression of PD-L1, as well as with the frequency of somatic mutations in the respective tumors. Patients with ATC / PDTC show high expression of PD-L1.

DETAILED DESCRIPTION:
Primary endpoint

1. Objective Response Ratio (ORR) [Time frame: prior to study completion, average 3 years]

   * Evaluate the effectiveness of a combination of a PD-1 inhibitor (pembrolizumab) with a multikinase inhibitor (lenvatinib) using an objective response rate (ORR) in poorly differentiated or anaplastic thyroid cancer at 12 weeks and 24 weeks after starting treatment.
   * Evaluate the efficacy of the investigator's choice of chemotherapy plus PD-1 inhibitor (pembrolizumab) using an objective response rate (ORR) in poorly differentiated or anaplastic thyroid cancer at 12 weeks and 24 weeks after initiation of treatment. Includes patients with a confirmed partial (PR) and complete response (CR) as the best response according to RECIST v 1.1.
2. Overall survival at 6 months in the pembrolizumab and lenvatinib cohort [Time frame: 6 months]

Secondary endpoints

1. Safety Profile (Number / Severity of Serious Adverse Events, SAEs) [Timeline: SAEs will be reported in the clinical trial within 6 months of the end of the study]
2. Duration of Response (DoR) [Time frame: from date of first documented clinical response (PR, CR) to date of first documented progression, date of death from any cause or patient failure, whichever comes first, is estimated to be 36 months]
3. Progression-Free Survival (PFS) [Time frame: from date of enrollment to date of first documented progression, date of death from any cause or patient failure, whichever is earlier, up to 36 months]
4. Overall Survival (OS) [Time frame: from the date of enrollment to the date of death from any cause or patient failure, whichever comes first, estimated up to 36 months]

Study design Prospective interventional two-cohort non-comparative single-center study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥ 18 years of age.
2. Willingness to participate in the research by signing an informed consent form approved by the research ethics committee.
3. ECOG status 0 or 1 or 2.
4. Measurable disease according to RECIST 1.1, as defined by the investigator.
5. Patients with a histologically confirmed disease (according to the pathologist's report) that meets one of the following criteria (according to the 2010 WHO classification):

   Poorly differentiated iodine-refractory thyroid tumors in the first line or after switching to chemotherapy or investigational drugs or anaplastic thyroid cancer in the first line or after switching to chemotherapy or investigational drugs. The primary tumor may or may not be removed, but the risk of aerodigestive compression or bleeding should be excluded.
6. Radioactive iodine resistant disease (RAI), which is defined by one or more of the following criteria:

   * One or more measurable lesions that do not show RAI uptake.
   * One or more measurable lesions progressing on RECIST 1.1 = <14 months prior RAI therapy
   * One or more measurable lesions are present after a cumulative dose of RAI> = 600 mCi
   * One or more measurable lesions that are F-18 fludeoxyglucose (FDG) -avid (> 5 standardized absorbance value [SUV]) if positron emission tomography (PET) / CT is performed; these lesions can also be RAI-active
7. Patients with inoperable locally advanced disease or metastases. Patients who do not want to undergo surgery or radiation are also eligible. Patients with the BRAFV600E mutation who are unable to take FDA-approved drugs, dabrafenib / trametinib, or established progression with therapy are eligible for study treatment if documented.
8. Ability to collect samples, including blood and tumors, for translational studies.
9. Weight over 30 kg.
10. Recovery from toxicity associated with any prior treatment to grade ≤ 1, unless adverse events (AEs) are clinically significant and / or are stable with maintenance therapy.
11. Ability to swallow pills or have a gastrostomy.
12. Normal organ and bone marrow function as defined below (obtained = <30 days prior to study entry):

    * Hemoglobin ≥ 9.0 g / dL.
    * Absolute neutrophil count (ANC)> 1500 per mm.
    * Platelet count ≥ 100,000 per mm.
    * Serum bilirubin ≤ 1.5 times the upper limit of normal (ULN) if liver metastases are absent, in which case it should be ≤ 2X ULN. This does not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia, which is predominantly unconjugated in the absence of hemolysis or liver pathology); however, they will only be admitted after consulting their doctor.
    * Aspartate transaminase (AST) (SGOT) / alanine aminotransferase (ALT) (SGPT) ≤ 2.5x the institutional upper limit of normal, unless liver metastases are present, in which case it should be ≤ 3x ULN.
    * Measured creatinine clearance (CL)> 40 ml / min or Estimated creatinine clearance> 40 ml / min using the Cockcroft-Gault formula (Cockcroft and Gault, 1976) or 24-hour urine collection to determine creatinine clearance.
    * Albumin> = 2.5 mg / dL (received = <30 days prior to registration)
    * International normalized ratio (INR) or prothrombin time (PT) = <1.5 X ULN if the subject is not receiving anticoagulant therapy while PT or partial thromboplastin time (PTT) is within the therapeutic range of the intended use of anticoagulants
    * Activated partial thromboplastin time (APTT) = <1.5 x ULN if the subject is not receiving anticoagulant therapy while the PT or PTT is within the therapeutic range of the intended use of anticoagulants
13. Adequately controlled blood pressure with or without antihypertensive drugs, defined as blood pressure (BP) <150/90 mm Hg.
14. Female subjects of childbearing age (not surgically sterile or at least 2 years of age in postmenopausal women) must present a negative pregnancy test at screening and use a medically accepted double-barrier method of contraception (e.g. spermicide condom + IUD or cervical caps). In addition, they must agree to continue using this double-barrier method for the duration of the study and for 4 months after the end of study participation. Women will be considered postmenopausal if they have had amenorrhea within 12 months without an alternative medical cause. The following age requirements apply:

    1. Women under 50 are considered to be posttmenopausal if they have had amenorrhea for 12 months or more after stopping treatment with exogenous hormones, and if they have postmenpausal levels of luteinizing hormone and follicle-stimulating hormone or have undergone surgical sterilization (bilateral oophorectomy or hysterectomy)
    2. Women over 50 years of age will be considered postmenopausal if they have had amenorrhea for 12 months or more after stopping all exogenous hormonal drugs with the last menstrual period> 1 year ago, had a menopause caused by chemotherapy with the last menstrual period> 1 year ago, or underwent surgery sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
15. Men must agree to abstain from intercourse with a female partner or agree to use a double-barrier method of contraception (for example, a spermicide condom, in addition to the fact that their female partner is using some form of contraception, such as an intrauterine device (IUD) or cervical caps), at the time of the study and for 4 months after the end of participation in the study.
16. Patient willingness and ability to adhere to protocol throughout the study, including undergoing treatment, and availability for scheduled visits and examinations, including follow-up.

Exclusion Criteria:

1. The presence of a confirmed BRAF mutation.
2. Concurrent participation in another clinical trial if it is not an observational (non-interventional) clinical trial or during the follow-up period of an interventional trial
3. Pretreatment with any immune checkpoint inhibitor therapy (eg anti-CTLA4, -PD-1 or -PD-L1).
4. Taking any type of low molecular weight kinase inhibitors (including the investigational kinase inhibitor) for 2 weeks or 5 half-lives of the agent, whichever is greater.
5. Receiving any type of anti-tumor antibodies (including test antibodies) or systemic chemotherapy within 2 weeks before starting treatment.
6. Current or previous use of immunosuppressants within 2 weeks prior to the first dose of study drugs, with the exception of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses that should not exceed 10 mg / day of prednisone or an equivalent corticosteroid.
7. Active or previously documented autoimmune disease within the past 2 years. Note: Patients with vitiligo, Graves' disease or psoriasis who do not require systemic treatment (within the last 2 years) are not excluded.
8. Active or previously documented inflammatory bowel disease (eg Crohn's disease and ulcerative colitis).
9. History of allogeneic organ transplantation.
10. Subjects diagnosed with immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 28 days prior to the first dose of study treatment.
11. Received radiation therapy for bone metastases within 2 weeks or any other radiation therapy within 4 weeks prior to enrollment. Subjects with clinically significant ongoing complications from previous radiation therapy that have not completely resolved are not eligible for the study (eg, radiation esophagitis or other internal inflammation).
12. Presence of metastases in the brain or epidural disease of the skull without adequate treatment with radiation therapy and / or surgery (including radiosurgery). Eligible patients should be neurologically asymptomatic and not receive corticosteroid medications during investigational treatment.
13. Concomitant therapy with oral anticoagulants (eg warfarin, direct thrombin and factor Xa inhibitors) or platelet inhibitors (eg clopidogrel), with the exception of the following approved anticoagulants:

    * Low-dose aspirin for cardioprotection (in accordance with current local guidelines) and low-dose low molecular weight heparins (LMWH).
    * Anticoagulant therapy with therapeutic doses of LMWH in subjects without known brain metastases who received a dose of LMWH for at least 6 weeks prior to enrollment and who had no clinically significant hemorrhagic complications from the anticoagulation regimen or tumor.
14. Subject has an uncontrolled, serious underlying medical condition or recent illness, including but not limited to the following conditions:

    A) Cardiovascular diseases:
    * Congestive heart failure, grade 3 or 4 as defined by the New York Heart Association, unstable angina, and severe cardiac arrhythmias.
    * Uncontrolled hypertension, defined as sustained blood pressure> 150 mm Hg. Systolic or diastolic> 100 mmHg
    * Stroke, including transient ischemic attack (TIA), myocardial infarction, other ischemic events or thromboembolic event, such as deep vein thrombosis (DVT) and pulmonary embolism) within 6 months prior to inclusion. Subjects with a later diagnosis of DVT are eligible if they are stable, asymptomatic, and have received LMWH for at least 6 weeks prior to study treatment.

    B) Gastrointestinal disorders (eg malabsorption syndrome or obstruction of the gastric outlet), including those associated with a high risk of perforation or fistula formation:
    * Active peptic ulcer disease, inflammatory bowel disease, ulcerative colitis, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis or acute obstruction of the pancreas or bile ducts, or obstruction of the gastric outlet.
    * Abdominal fistula, gastrointestinal perforation, bowel obstruction, or intra-abdominal abscess within 6 months prior to inclusion. Note: Complete healing of the intra-abdominal abscess must be confirmed before starting treatment.

    C) Clinically significant vomiting or hemoptysis> 0.5 teaspoon (> 2.5 ml) of red blood or other significant bleeding in history within 3 months prior to treatment.

    D) Interstitial lung lesions or known manifestations of endobronchial disease. F) Lesions invading the main pulmonary blood vessels.

    F) Other clinically significant disorders such as:
    * An active infection requiring systemic treatment, infection with human immunodeficiency virus or disease associated with acquired immunodeficiency syndrome, or chronic infection with hepatitis B or C.
    * Serious non-healing wound / ulcer / bone fracture.
    * Moderate or severe liver failure (Child-Pugh B or C).
    * The need for hemodialysis or peritoneal dialysis.
    * Uncontrolled diabetes mellitus.
    * History of solid organ transplantation.
15. Major surgery (such as gastrointestinal surgery and removal or biopsy of brain metastases) within 8 weeks prior to inclusion. Complete wound healing from major surgery should occur 4 weeks before the study treatment, and after minor surgery (eg, simple excision, tooth extraction) at least 10 days before the study treatment. Patients with clinically significant ongoing complications from prior surgery are not eligible.
16. Adjusted QT interval calculated by Fridericia formula (QTcf)> 500 ms for 28 days prior to study treatment.

    Note: If a single ECG displays a QTCf with an absolute value> 500 ms, two additional ECGs at approximately 3 min intervals must be performed within 30 minutes of the initial ECG, and the average of these three consecutive results will be used to assess eligibility for study participation.
17. Pregnant (test must be done no later than 7 days before the start of the study) or lactating mothers.
18. Received any live vaccine = <30 days prior to study initiation.
19. Inability to swallow pills and lack of gastrostomy.
20. Previously identified allergy or hypersensitivity to the components of the investigational dosage forms.
21. Diagnosis of other malignant neoplasm within 3 years prior to study treatment, with the exception of superficial skin cancer or localized low-grade tumors that are considered cured and untreated by systemic therapy.
22. ADDITIONAL EXCLUSION CRITERION FOR COHORT 1 (pembrolizumab + lenvatinib): The presence of invasion (germination) of the tumor into the major great vessels or the presence of clinically significant blood clots in the arteries or veins.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2023-12-28 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | prior to study completion, average 3 years
  ORR will be calculated as the number of patients with an observed response divided by the number of patients included in the study. A two-sided confidence interval will be calculated at 80% (in accordance with the specified α) and 95% (for comparison with the literature).
Overall survival at 6 months in cohort Lenvatinib+Pembrolizumab | 6 months
  Overall survival is defined as the time from the date of initiation of treatment to death from any cause that will be assessed using the Kaplan-Meier method.

SECONDARY OUTCOMES:
Safety Profile (Number / Severity of Serious Adverse Events, SAEs) | SAEs will be reported in the clinical trial within 6 months of the end of the study
  Number of serious adverse events classified by severity as assessed by CTCAE v4.0
Duration of Response (DoR) | from date of first documented clinical response (PR, CR) to date of first documented progression, date of death from any cause or patient failure, whichever comes first, is estimated to be 36 months
  Time from the date of the first documented CR or PR to the first documented progression or death due to cancer. DoR will be determined based on tumor score (RECIST criteria version 1.1).
Progression-Free Survival (PFS) | from date of enrollment to date of first documented progression, date of death from any cause or patient failure, whichever is earlier, up to 36 months
  Median progression-free survival (mPFS) is defined as the time from the date of inclusion to the date of the first documented progression of disease or death from any cause, whichever occurs first. PFS will be determined based on the tumor score (RECIST criteria version 1.1).
Overall Survival (OS) | from the date of enrollment to the date of death from any cause or patient failure, whichever comes first, estimated up to 36 months
  Mean overall survival (mOS) is calculated as the time from the date of inclusion to the date of death for any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Yuliya Mikheeva, M.D., Ph.D., Principal Investigator — Saint-Petersburg State University (SPSU) N.I.Pirogov Clinic of High Medical Technologies
Locations (1):
- Saint-Petersburg State University (SPSU) N.I.Pirogov Clinic of High Medical Technologies, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No